CLINICAL TRIAL: NCT07123558
Title: Anal Cancer Prevention in High-Risk Categories of Men Who Have Sex With Men - A Danish Prospective Study
Brief Title: Anal Cancer Prevention in High-Risk Categories of Men Who Have Sex With Men
Acronym: DACaP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Vejle Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helle Kiellberg Larsen, consultant, Bispebjerg Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: S-20240079; 2024-0039 (Other Grant/Funding Number: The Capital Region of Denmark Research Foundation); No grant number (Other Grant/Funding Number: Bispebjerg and Frederiksberg Hospital Research Fund); KC23-00598 (Other Grant/Funding Number: The Danish Cancer Society Prevention Lab); KC25-01568 (Other Grant/Funding Number: The Danish Cancer Society Knæk Cancer)
Record Dates: First submitted 2025-07-11; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anal HSIL; Anal AIN3; Anal HPV Infection
Keywords: anal HSIL; HIV infection; MSM; anal HPV infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: a prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High resolution anoscopy (Other): MSM with or without HIV infection will be examined with high-resolution anoscopy for anal HSIL lesions and anal warts additionally with anal swabs for HPV and cytology and dual stain cytology, comparing the two groups over time (baseline and 1 year follow up visit)
  Interventions: Diagnostic Test: High resolution anoscopy

INTERVENTIONS:
Diagnostic Test: High resolution anoscopy — to study biomarkers for anal cancer screening
  Other Names: Anal cancer screening

SUMMARY:
The incidence of anal cancer is increasing, particularly among high-risk groups such as men who have sex with men (MSM), especially those living with HIV. The lack of comprehensive screening programs results in delayed diagnosis and higher mortality.

This project aims to establish a screening program for anal cancer in high-risk populations, with a specific focus on those most at risk. Using a prospective study design, the project will assess the effectiveness of early detection and prevention strategies to potentially reduce cancer incidence and improve survival rates. If an HPV-based screening method proves effective, it would serve as a potential implemention for high-risk groups in Denmark, further enhancing early detection and prevention efforts.

This study represents the first large-scale, prospective screening initiative for anal cancer in Denmark,specifically targeting MSM. It introduces a novel approach to cancer prevention in this population by building on research in other cancers and adapting it to anal cancer and its specific risk factors.

The project is a collaboration between clinical practitioners and academic researchers, ensuring that practical clinical insights guide the research and that research findings are rapidly translated into clinical practice. This partnership will enhance both the quality of the research and its direct application in healthcare.

The project is expected to lead to earlier diagnosis of anal cancer, reduced morbidity and mortality among high-risk populations, and the establishment of a screening model that can be applied nationwide. This could significantly reduce the overall healthcare burden associated with late-stage anal cancer and improve patient outcomes across Denmark.

DETAILED DESCRIPTION:
Background:

Anal cancer can potentially be prevented by introducing screening in Denmark. This is in line with the existing cervical cancer screening program available to Danish women aged 23 to 64 since the 1990s.

Anal squamous cell carcinoma (ASCC) is rare in the general population, with an incidence of 1-2 cases per 100,000 (1). In Denmark, approximately 160 new cases of ASCC are diagnosed annually (2), with around 50 fatalities each year. For comparison, there are about 300 cases of cervical cancer in Denmark and 90 related deaths annually. However, the incidence of ASCC has been significantly increasing over the past decades (3) and is expected to rise markedly in the coming years.

More than 80% of the anal cancers are ASCCs. ASCC are preceded by precancerous lesions, anal highgrade squamous intraepithelial lesions (HSIL) (4). ASCC and anal HSIL are caused by persistent infection with high-risk human papilloma virus (hrHPV), found in more than 90% of anal HSIL and ASCC cases, with HPV type 16 being the far most carcinogenic type (5, 6).

Certain populations, including people with HIV and men who have sex with men (MSM), have a significantly higher risk of ASCC and its precancerous lesions (7-10). MSM with HIV constitutes the highest risk of anal cancer with an incidence of anal cancer >70/100,000(1) which is more than 50-times the risk of the general population (10). Pre-exposure prophylaxis (PrEP) is the use of antiviral drugs to protect high-risk populations from acquiring human immunodeficiency virus (HIV) (11). In Denmark, this treatment is offered to people at increased risk of HIV, with the majority being HIV-negative MSM who are engage in high-risk behaviors, such as having multiple sex partners and unprotected anal intercourse and having had recent sexually transmitted infections (STIs) (12).

A recent Danish registry-based study showed a 5-year risk of anal cancer following anal HSIL of 14.1% among people with HIV compared with 3.2% among HIV negative individuals (7). A significant proportion of MSM harbor anal hrHPV. The reported prevalence of anal hrHPV among MSM with HIV and HIV negative MSM on preexposure prophylaxis (MSMonPrEP) is 74-85% (13, 14). The 5-year survival rate after anal cancer is 80% for patients with tumor size < 2 cm and 45-65% with tumor size >2 cm(15). A Danish registry-based study found that only one third of patients diagnosed with ASCC were diagnosed in a local stage, while 6.5% exhibited distant metastasis (16). It is therefore pivotal to prevent the development of ASCC or to diagnose in an early stage.

Therefore, with a targeted effort among high-risk populations in Denmark by examination for precancerous lesions in the anal canal and perianal area most cases of anal cancer could be prevented or detected early, thereby decreasing the risk of cancer spreading and associated mortality. HPV vaccination is expected to be another major long-term solution to ASCC prevention in both men and women(17-19). However, the full impact will not be seen for decades, and many high-risk individuals are already infected with hrHPV, making the vaccine's effectiveness in this group unclear. The ANCOR study (20), a large American multicenter study including more than 4,000 people living with HIV and with histologically confirmed anal HSIL, compared active monitoring with active treatment of anal HSIL using high-resolution anoscopy (HRA). The study found a 57% reduction in risk of progression to ASCC in the treatment arm. The cumulative incidence of progression to anal cancer at 48 months was 0.9% in the treatment group and 1.8% in the active-monitoring group. The risk of progression from anal/perianal HSIL to ASCC increased with size and extent of the lesions. Therefore, missed opportunities likely exist in preventing anal cancer progression from treatable precursor lesions. Consequently, there is an unmet need to clarify whether screening and treatment of anal HSIL in Danish risk-populations is beneficial and to evaluate the necessity of implementing national screening protocols for anal cancer among high-risk populations, especially MSM and people with HIV. Systematic data collection within the Danish population is crucial to identify the high-risk groups that should be offered screening interventions and to test the effectiveness of screening methods before proposing suitable national screening algorithms. With the introduction of a new method in the form of DNA methylation analysis and plasma HPV analysis (pHPV), we hope to predict those individuals who should be offered closer follow-up in the long term, thereby limiting overtreatment/over-testing and all that this entails.

Screening Modalities Since the 1990s, a secondary prevention tool for anal cancer has emerged: high-resolution anoscopy (HRA). This procedure is akin to colposcopy for the cervix, as both HSIL lesions in these areas typically arise in the transformation zone where the columnar and squamous epithelium meets(21, 22).

In November 2023, the International Anal Neoplasia Society (IANS) released their consensus guidelines on anal cancer screening for high-risk groups(10). Individuals with a more than 10-fold increased risk of anal cancer are advised to be screened. This aligns with the European guidelines for HIV cancer screening from the European AIDS Clinical Society (EACS)(23). Despite these recommendations, there are currently no Danish guidelines for screening for anal ASCC in high-risk populations.

Screening Tests Anal cytology, HPV testing (genotyping), and hrHPV-cytology co-testing are all currently used strategies for anal cancer screening with acceptable results. hrHPV alone may also be used. Triage using hrHPV testing can reduce the need for referral to HRA. As both sensitivity and specificity of anal cytology is limited, co-testing for anal hrHPV has shown to increase the sensitivity of anal cytology, but the high prevalence of hrHPV in MSM with HIV compromise sensitivity(22). There is a need for prognostic markers to improve screening algorithms for HRA referral. Promising biomarkers, including p16/Ki 67 dual staining, and DNA methylation analysis, are demonstrating potential for future triage testing approaches(5, 24-30). Circulating plasma HPV (pHPV) is being evaluated as a biomarker in a phase III study (NOAC9)(31) for early treatment failure or recurrence in anal cancer patients, showing promising preliminary results. Recent technological advances have enabled the sensitive and reliable identification and quantification of low copy number HPV gene expression in blood. This project will be the first to investigate whether circulating pHPV in participants with biopsy confirmed anal HSIL can serve as a future biomarker in anal cancer screening.

AIM:

The overall aim in a prospective cohort study is:

1. To investigate the use of HPV-based anal cancer screening for early detection of anal cancer and its precancer lesions in two Danish high-risk populations: MSM with HIV and MSMonPrEP
2. To examine the diagnostic potential of biomarkers (p16/ki67 dual stain cytology, DNA methylation analysis and pHPV).

Additionally, the study aims to:

1. Assess the prevalence, incidence, persistence and risk of anal hrHPV in two Danish high-risk population of MSM with HIV and MSMonPrEP
2. To evaluate the diagnostic accuracy and feasibility of HPV analysis on self-collected anal samples compared to HPV analysis on professionally collected cell samples
3. To investigate the diagnostic potential of pHPV (blood test) as a future biomarker for anal HSIL
4. Assess the prevalence, incidence, and risk of anogenital warts and anal HSIL in a Danish population of MSM with HIV compared with MSMonPrEP triaged to high-resolution anoscopy (HRA).
5. Identify risk factors for anal hrHPV, anal HSIL, and intra- and perianal warts in Danish MSM with HIV and MSMonPrEP, including lifestyle factors, sexual behavior, sexually transmitted infections (STIs), and the CD4/CD8 ratio.
6. Evaluate the study participants experiences with the screening examination, and the impact it has on them through a questionnaire or individual interviews.
7. Evaluate the socio-economic perspective of implementing this screening (in collaboration with the Danish Center of Health Economics, SDU and Sisse Njor, Professor of population-based cancer screening programmes. Department of Regional Health Research, SDU and Lillebaelt Hospital)

Materials and Methods:

The study is designed as a prospective observational multicenter study. The investigators aim to include 350 MSM with HIV from the Department of Infectious Diseases, Aarhus University Hospital, Copenhagen University Hospital, Hvidovre Hospital, and Copenhagen University Hospital, Rigshospitalet, where they attend regular HIV follow-up (typically one or twice annually), as well as from the Clinic for Sexually Transmitted Infections (STI) at Copenhagen University Hospital, Bispebjerg Hospital, where they undergo STI screening. Additionally, the investigators will include a control group of 350 HIV negative MSMonPrEP from the same departments. Participants will be asked to participate when they are attending for regular outpatient follow-up appointments or STI screening.

Questionnaire All participants will be asked to complete a lifestyle and sexual behavior questionnaire at time of inclusion and after 1-year follow-up visit.

Anal samples for Anal Cytology, Biomarkers, and DNA Methylation Analysis The study includes HPV-based anal cancer screening. Anal samples for HPV will be performed by the two High-resolution anoscopy providers at baseline and at 1-year follow-up. Additionally, 80 participants, equivalent to 10-15%, will be asked to perform an anal self-test for HPV analysis at baseline and at 1-year follow-up.

The anal liquid-based cytology is collected using a standard cytobrush, which is inserted into the anal canal rotating while withdrawing. Histologically confirmed HSIL, will have methylation analysis performed. In addition, a blood sample will be collected from participants with biopsy-confirmed anal HSIL to analyze circulating plasma HPV (pHPV blood sample). The blood samples will be analyzed at Department of Pathology, Vejle Hospital. Anal samples for HPV testing, cytology, and p16/Ki67 dual stain cytology analysis will be analyzed at the Department of Pathology, Vejle Hospital and DNA methylation at Randers Hospital.

HPV genotyping will be conducted using the INNO-LiPA test (Fujirebio) to detect DNA from 32 HPV types. This includes 13 high-risk types. Through HPV genotyping, participants will be tested for the persistence of specific genotypes. Anal samples will be tested consecutively, with results communicated to participants.

High-resolution anoscopy All participants will have high-resolution anoscopy (HRA) performed. HRA differs from standard anoscopy by the application of acetic acid 5% and iodine-based Lugol's solution, and visualization under magnification of lesions that would otherwise be invisible. During the procedure the anal canal and the perianal area will be examined for warts and precancerous lesions. The procedure is preceded by a digital anal rectal examination using a water-soluble lubricant mixed with 2-5% lidocaine gel or cream. The anoscope is inserted and a Q-tip wrapped in gauze soaked in 5% acetic acid is inserted and left for 2 minutes, the whole transformation zone is visualized during magnification of a colposcope. The perianal area is likewise visualized after acetic acid application for 2 minutes. Lesions indicative for HSIL or warts will be biopsied and send for histopathological examination at a highly specialized department of Pathology. The biopsies will be taken using biopsy forceps. Digital photos will be taken for documentation during HRA using a digital camara connected to the colposcope.

Participants with biopsy proven anal HSIL by HRA will be offered treatment according to gold standard by either topical (aldara, topical 5-flourouracil or topical cidofovir 2%) or ablative treatment (electrocautery). After treatment the participants will be followed every 6 months with HRA until no signs of anal HSIL and then continue study flow as scheduled.

Statistical analyses:

The prevalence and incidence of anal HPV infection and HSIL will be calculated with descriptive statistics. Prevalence will be calculated overall and separately for low- and high-risk HPV types.

Comparisons between MSM with HIV and MSMonPrEP will be analyzed using chi-squared test and regression models. Associations between outcomes (anal HPV infection, anal HSIL, anal warts) and exposure variables will be evaluated by means of regression models, e.g. Cox regression models or logistic regression models providing hazard ratios (HRs) or odds ratios (Ors), respectively, both with 95% confidence limits. Analyses will be performed overall and separately for the MSM with HIV and MSMonPrEP.

Power calculation and sample size The study is designed to have sufficient statistical power to determine a difference in anal hrHPV, anal warts, and anal HSIL prevalence and incidence in MSM with HIV and MSMonPrEP. The power calculation was performed using a two-sided likelihood ratio test with a significance level of ɑ=0.05. Based on data from the metaanalysis published in Lancet HIV (14), the investigators expect that approximately 74% of the MSM with HIV and 84% of the MSMonPrEP will have incident anal hrHPV infection at the one-year follow-up visit, yielding a power of 88.6%. Additionally, with an expected HSIL prevalence of 22.4% in MSM with HIV and 11.3% in MSMonPrEP (13), and a sample size of 350 in each group, the power to detect the expected difference is 97.6%.

Ethical requirements:

The study will be conducted in accordance with the Helsinki Declaration (2002) after approval by the Regional Scientific Ethical Committee. A RedCap database will be established for the study. All participants will be throughly informed about the purpose and content of the study.

ELIGIBILITY:
Inclusion Criteria:

* MSM with HIV
* HIV-negative MSMonPrEP
* Age >=35 years
* Written and orally informed consent in English or Danish

Exclusion criteria

* Previous anal cancer
* Rectum extirpation (of any cause)
* Unwilling to have HRA performed
* Inflammatory bowel disease
* Inability and unwillingness to give informed consent
* Other known immunosuppressive disorder than HIV
* No sex with men

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Anal HSIL prevalence and incidence | 1 year
  Anal HSIL defined as the result of findings on HRA confirmed histologically at baseline and 1-year follow-up in HIV positive MSM compared to MSM on PrEP
Anal high-risk HPV infection | 1-2 years
  Anal HPV infection defined as the result of anal HPV test, including prevalence, incidence, and persistent infections.MSM living with HIV compared to MSM on PrEP

SECONDARY OUTCOMES:
The diagnostic potential of biomarkers (p16/ki67 dual stain cytology, DNA methylation analysis and pHPV). | 1-2 years
  Performance of HPV test, anal cytology, and biomarkers (p16/Ki-67 dual stain, DNA methylation analysis, pHPV), sensitivities and specificities to predict anal HSIL.
Anal warts prevalence and incidence | 1-2 year
  Anal and perianal warts defined as findings on HRA confirmed histologically inMSM living with HIV compared to MSM on PrEP

OTHER OUTCOMES:
Performance of HPV self-test compared to professional collected anal samples | 1 year
  The diagnostic accuracy and feasibility of HPV analysis on self-collected anal samples compared to HPV analysis on professionally collected cell samples for 15% of the participants

REFERENCES:
- [Background] Group DAC. NOAC 9 - A Phase III Randomized Nordic Anal Cancer Group Study on Circu-lating Tumor DNA guided Follow-Up. https://wwwdcccdk/english/projectsandnetwork/noac-9---a-phase-iiirandomized-nordic-anal-cancer-group-study-on-circulating-tumor-dna-guided-follow-up/.
- [Background] van der Zee RP, van Noesel CJM, Martin I, Ter Braak TJ, Heideman DAM, de Vries HJC, Prins JM, Steenbergen RDM. DNA methylation markers have universal prognostic value for anal cancer risk in HIV-negative and HIV-positive individuals. Mol Oncol. 2021 Nov;15(11):3024-3036. doi: 10.1002/1878-0261.12926. Epub 2021 Mar 16. PMID 33580586
- [Background] Swanson AA, Hartley C, Long ME, Chantigian PDM, Casey PM, Jenkins SM, Boerger AC, Binnicker MJ, Henry MR. Evaluation of high-risk human papillomavirus testing and anal cytology to detect high-grade anal intraepithelial neoplasia. J Am Soc Cytopathol. 2021 Jul-Aug;10(4):406-413. doi: 10.1016/j.jasc.2021.03.007. Epub 2021 Apr 6. PMID 33896747
- [Background] Goncalves JCN, Macedo ACL, Madeira K, Bavaresco DV, Dondossola ER, Grande AJ, da Rosa MI. Accuracy of Anal Cytology for Diagnostic of Precursor Lesions of Anal Cancer: Systematic Review and Meta-analysis. Dis Colon Rectum. 2019 Jan;62(1):112-120. doi: 10.1097/DCR.0000000000001231. PMID 30451747
- [Background] Hopp AM, Pant M, Sniedze S, Parsons LN, Hunt B, Giorgadze T. Correlation of anal cytology with follow-up histology and Human Papillomavirus genotyping: A 10-year experience from an academic medical center. Ann Diagn Pathol. 2021 Feb;50:151670. doi: 10.1016/j.anndiagpath.2020.151670. Epub 2020 Nov 20. PMID 33310590
- [Background] Patarapadungkit N, Khonhan P, Pisuttimarn P, Pientong C, Ekalaksananan T, Koonmee S. Human Papillomavirus Detection and Abnormal Anal Cytology in HIV-infected Patients Using p16/Ki-67 Dual-Staining. Asian Pac J Cancer Prev. 2020 Jul 1;21(7):2013-2019. doi: 10.31557/APJCP.2020.21.7.2013. PMID 32711427
- [Background] Clarke MA, Cheung LC, Lorey T, Hare B, Landy R, Tokugawa D, Gage JC, Darragh TM, Castle PE, Wentzensen N. 5-Year Prospective Evaluation of Cytology, Human Papillomavirus Testing, and Biomarkers for Detection of Anal Precancer in Human Immunodeficiency Virus-Positive Men Who Have Sex With Men. Clin Infect Dis. 2019 Aug 1;69(4):631-638. doi: 10.1093/cid/ciy970. PMID 30418518
- [Background] Macedo AC, Grande AJ, Figueiredo T, Colonetti T, Goncalves JC, Testoni E, da Rosa MI. DNA high-risk HPV, mRNA HPV and P16 tests for diagnosis of anal cancer and precursor lesions: a systematic review and meta-analysis. EClinicalMedicine. 2023 Aug 11;62:102128. doi: 10.1016/j.eclinm.2023.102128. eCollection 2023 Aug. PMID 37588624
- [Background] European AIDS Clinical Society (EACS). https://www.eacsociety.org/guidelines/eacs-guidelines/ Assessed 17.04.2024
- [Background] Barroso LF, Stier EA, Hillman R, Palefsky J. Anal Cancer Screening and Prevention: Summary of Evidence Reviewed for the 2021 Centers for Disease Control and Prevention Sexually Transmitted Infection Guidelines. Clin Infect Dis. 2022 Apr 13;74(Suppl_2):S179-S192. doi: 10.1093/cid/ciac044. PMID 35416975
- [Background] Hillman RJ, Cuming T, Darragh T, Nathan M, Berry-Lawthorn M, Goldstone S, Law C, Palefsky J, Barroso LF, Stier EA, Bouchard C, Almada J, Jay N. 2016 IANS International Guidelines for Practice Standards in the Detection of Anal Cancer Precursors. J Low Genit Tract Dis. 2016 Oct;20(4):283-91. doi: 10.1097/LGT.0000000000000256. PMID 27561134
- [Background] Palefsky JM, Lee JY, Jay N, Goldstone SE, Darragh TM, Dunlevy HA, Rosa-Cunha I, Arons A, Pugliese JC, Vena D, Sparano JA, Wilkin TJ, Bucher G, Stier EA, Tirado Gomez M, Flowers L, Barroso LF, Mitsuyasu RT, Lensing SY, Logan J, Aboulafia DM, Schouten JT, de la Ossa J, Levine R, Korman JD, Hagensee M, Atkinson TM, Einstein MH, Cracchiolo BM, Wiley D, Ellsworth GB, Brickman C, Berry-Lawhorn JM; ANCHOR Investigators Group. Treatment of Anal High-Grade Squamous Intraepithelial Lesions to Prevent Anal Cancer. N Engl J Med. 2022 Jun 16;386(24):2273-2282. doi: 10.1056/NEJMoa2201048. PMID 35704479
- [Background] Baandrup L, Maltesen T, Dehlendorff C, Kjaer SK. Human papillomavirus vaccination and anal high-grade precancerous lesions and cancer-a real-world effectiveness study. J Natl Cancer Inst. 2024 Feb 8;116(2):283-287. doi: 10.1093/jnci/djad189. PMID 37718496
- [Background] Palefsky JM, Lensing SY, Belzer M, Lee J, Gaur AH, Mayer K, Futterman D, Stier EA, Paul ME, Chiao EY, Reirden D, Goldstone SE, Tirado M, Cachay ER, Barroso LF, Da Costa M, Darragh TM, Rudy BJ, Wilson CM, Kahn JA. High Prevalence of Anal High-Grade Squamous Intraepithelial Lesions, and Prevention Through Human Papillomavirus Vaccination, in Young Men Who Have Sex With Men Living With Human Immunodeficiency Virus. Clin Infect Dis. 2021 Oct 20;73(8):1388-1396. doi: 10.1093/cid/ciab434. PMID 33991185
- [Background] Goldstone SE, Giuliano AR, Palefsky JM, Lazcano-Ponce E, Penny ME, Cabello RE, Moreira ED Jr, Baraldi E, Jessen H, Ferenczy A, Kurman R, Ronnett BM, Stoler MH, Bautista O, Das R, Group T, Luxembourg A, Zhou HJ, Saah A. Efficacy, immunogenicity, and safety of a quadrivalent HPV vaccine in men: results of an open-label, long-term extension of a randomised, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2022 Mar;22(3):413-425. doi: 10.1016/S1473-3099(21)00327-3. Epub 2021 Nov 12. PMID 34780705
- [Background] Urbute A, Munk C, Sand FL, Belmonte F, Kjaer SK. Trends in incidence and survival from anal cancer and incidence of high-grade anal intraepithelial neoplasia in Denmark. Cancer Epidemiol. 2022 Apr;77:102099. doi: 10.1016/j.canep.2022.102099. Epub 2022 Jan 13. PMID 35033922
- [Background] Hillman RJ, Berry-Lawhorn JM, Ong JJ, Cuming T, Nathan M, Goldstone S, Richel O, Barrosso LF, Darragh TM, Law C, Bouchard C, Stier EA, Palefsky JM, Jay N; International Anal Neoplasia Society. International Anal Neoplasia Society Guidelines for the Practice of Digital Anal Rectal Examination. J Low Genit Tract Dis. 2019 Apr;23(2):138-146. doi: 10.1097/LGT.0000000000000458. PMID 30907777
- [Background] Cotte L, Veyer D, Charreau I, Pere H, Cua E, Carette D, Chas J, Capitant C, Chidiac C, Flejou JF, Fouere S, Heard I, Meyer L, Puech J, Tremblay C, Delaugerre C, Molina JM. Prevalence and Incidence of Human Papillomavirus Infection in Men Having Sex With Men Enrolled in a Pre-exposure Prophylaxis Study: A Sub-study of the Agence Nationale de Recherches sur le SIDA et les Hepatites Virales "Intervention Preventive de l'Exposition aux Risques avec et pour les hommes Gays" Trial. Clin Infect Dis. 2021 Jan 23;72(1):41-49. doi: 10.1093/cid/ciaa002. PMID 31907521
- [Background] Wei F, Gaisa MM, D'Souza G, Xia N, Giuliano AR, Hawes SE, Gao L, Cheng SH, Dona MG, Goldstone SE, Schim van der Loeff MF, Neukam K, Meites E, Poynten IM, Dai J, Combes JD, Wieland U, Burgos J, Wilkin TJ, Hernandez AL, Iribarren Diaz M, Hidalgo-Tenorio C, Valencia Arredondo M, Nyitray AG, Wentzensen N, Chow EP, Smelov V, Nowak RG, Phanuphak N, Woo YL, Choi Y, Hu Y, Schofield AM, Woestenberg PJ, Chikandiwa AT, Hickey AC, de Pokomandy A, Murenzi G, Pere H, Del Pino M, Ortiz AP, Charnot-Katsikas A, Liu X, Chariyalertsak S, Strong C, Ong JJ, Yunihastuti E, Etienney I, Ferre VM, Zou H, Segondy M, Chinyowa S, Alberts CJ, Clifford GM. Epidemiology of anal human papillomavirus infection and high-grade squamous intraepithelial lesions in 29 900 men according to HIV status, sexuality, and age: a collaborative pooled analysis of 64 studies. Lancet HIV. 2021 Sep;8(9):e531-e543. doi: 10.1016/S2352-3018(21)00108-9. Epub 2021 Jul 30. PMID 34339628
- [Background] Engsig FN, Kronborg G. Pre-exposure prophylaxis against HIV infection. Ugeskr Laeger. 2024 May 6;186(19):V10230672. doi: 10.61409/V10230672. Danish. PMID 38808765
- [Background] McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, Sullivan AK, Clarke A, Reeves I, Schembri G, Mackie N, Bowman C, Lacey CJ, Apea V, Brady M, Fox J, Taylor S, Antonucci S, Khoo SH, Rooney J, Nardone A, Fisher M, McOwan A, Phillips AN, Johnson AM, Gazzard B, Gill ON. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet. 2016 Jan 2;387(10013):53-60. doi: 10.1016/S0140-6736(15)00056-2. Epub 2015 Sep 9. PMID 26364263
- [Background] Stier EA, Clarke MA, Deshmukh AA, Wentzensen N, Liu Y, Poynten IM, Cavallari EN, Fink V, Barroso LF, Clifford GM, Cuming T, Goldstone SE, Hillman RJ, Rosa-Cunha I, La Rosa L, Palefsky JM, Plotzker R, Roberts JM, Jay N. International Anal Neoplasia Society's consensus guidelines for anal cancer screening. Int J Cancer. 2024 May 15;154(10):1694-1702. doi: 10.1002/ijc.34850. Epub 2024 Jan 31. PMID 38297406
- [Background] Sunesen KG, Norgaard M, Thorlacius-Ussing O, Laurberg S. Immunosuppressive disorders and risk of anal squamous cell carcinoma: a nationwide cohort study in Denmark, 1978-2005. Int J Cancer. 2010 Aug 1;127(3):675-84. doi: 10.1002/ijc.25080. PMID 19960431
- [Background] Reinholdt K, Thomsen LT, Dehlendorff C, Larsen HK, Sorensen SS, Haedersdal M, Kjaer SK. Human papillomavirus-related anogenital premalignancies and cancer in renal transplant recipients: A Danish nationwide, registry-based cohort study. Int J Cancer. 2020 May 1;146(9):2413-2422. doi: 10.1002/ijc.32565. Epub 2019 Aug 2. PMID 31291470
- [Background] Faber MT, Frederiksen K, Palefsky JM, Kjaer SK. Risk of Anal Cancer Following Benign Anal Disease and Anal Cancer Precursor Lesions: A Danish Nationwide Cohort Study. Cancer Epidemiol Biomarkers Prev. 2020 Jan;29(1):185-192. doi: 10.1158/1055-9965.EPI-19-0601. Epub 2019 Oct 9. PMID 31597665
- [Background] Lin C, Franceschi S, Clifford GM. Human papillomavirus types from infection to cancer in the anus, according to sex and HIV status: a systematic review and meta-analysis. Lancet Infect Dis. 2018 Feb;18(2):198-206. doi: 10.1016/S1473-3099(17)30653-9. Epub 2017 Nov 17. PMID 29158102
- [Background] Chowdhury S, Darragh TM, Berry-Lawhorn JM, Isaguliants MG, Vonsky MS, Hilton JF, Lazar AA, Palefsky JM. HPV Type Distribution in Benign, High-Grade Squamous Intraepithelial Lesions and Squamous Cell Cancers of the Anus by HIV Status. Cancers (Basel). 2023 Jan 20;15(3):660. doi: 10.3390/cancers15030660. PMID 36765617
- [Background] Darragh TM, Colgan TJ, Cox JT, Heller DS, Henry MR, Luff RD, McCalmont T, Nayar R, Palefsky JM, Stoler MH, Wilkinson EJ, Zaino RJ, Wilbur DC; Members of LAST Project Work Groups. The Lower Anogenital Squamous Terminology Standardization Project for HPV-Associated Lesions: background and consensus recommendations from the College of American Pathologists and the American Society for Colposcopy and Cervical Pathology. Arch Pathol Lab Med. 2012 Oct;136(10):1266-97. doi: 10.5858/arpa.LGT200570. Epub 2012 Jun 28. PMID 22742517
- [Background] Islami F, Ferlay J, Lortet-Tieulent J, Bray F, Jemal A. International trends in anal cancer incidence rates. Int J Epidemiol. 2017 Jun 1;46(3):924-938. doi: 10.1093/ije/dyw276. PMID 27789668
- [Background] Nordcan. https://gco.iarc.fr/media/nordcan/factsheets/93/en/countries/208/anus_and_anal_canal-105-denmark-208.pdf. Assessed February 22, 2024.
- [Background] Clifford GM, Georges D, Shiels MS, Engels EA, Albuquerque A, Poynten IM, de Pokomandy A, Easson AM, Stier EA. A meta-analysis of anal cancer incidence by risk group: Toward a unified anal cancer risk scale. Int J Cancer. 2021 Jan 1;148(1):38-47. doi: 10.1002/ijc.33185. Epub 2020 Jul 29. PMID 32621759